CLINICAL TRIAL: NCT06129929
Title: Using Kolb's Experiential Learning Program to Promote Nurse Effectiveness for Coping With Workplace Violence
Brief Title: Effectiveness of Using Jiu-Jitsu for Coping With Medical Violence in Healthcare Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hui-Hsun Chiang (Other)
Responsible Party: Sponsor-Investigator, Hui-Hsun Chiang, Professor, National Defense Medical Center, Taiwan
Organization: National Defense Medical Center, Taiwan (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BJJ
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Educational Problems; Workplace Violence; Nursing
Keywords: education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hospital Jujutsu Group, HJJ Group (Experimental): The intervention group participants who received the theoretical-based BJJ educational intervention.
  Interventions: Behavioral: Hospital Jujutsu Group, HJJ Group
- Traditional lecture Group (Active Comparator): The control group participants who received the traditional violence-prevention educational intervention.
  Interventions: Behavioral: Hospital Jujutsu Group, HJJ Group

INTERVENTIONS:
Behavioral: Hospital Jujutsu Group, HJJ Group — The aim of this study, procedures, methodology, and the subject's rights were well explained to the eligible nursing staff according to the informed consent form. Written informed consent was obtained from each participant before data collection.

SUMMARY:
Workplace violence in hospitals and other health care settings is a troublesome issue and has severe consequences for the entire health care system. In recent years, workplace violence has made a great threat to nurse assistants. Therefore, violence prevention education is a part of medical personnel's job responsibility. However, a theory-based violence prevention education program for healthcare settings was limited. The aim of the study is to investigate the effects of experiential learning theory-based medical jujitsu training on perception on violence, attitude on violence, self-efficacy, and turnover intention among nurse assistants

ELIGIBILITY:
Inclusion Criteria:

* Licensed healthcare professionals

Exclusion Criteria:

* Non-licensed healthcare professionals

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Self efficacy | pre and post intervention
  Self efficacy was measured by the General Self-Efficacy Scale (GSES). The scale was consists of 10 items, rating from 1 (Not at all true) to 4 (Exactly true). The sum of scores ranged from 10 to 40, with a higher score indicating a higher level of self efficacy.

SECONDARY OUTCOMES:
Perception of Aggression | pre and post intervention
  Perception of aggression was measured by the Perception of Aggression Scale (POAS). The scale was consists of 18 items, rating from 1 (Strongly disagree) to 5 (Strongly agree). The sum of scores ranged from 18 to 90, with a higher score indicating a more positive view and higher tolerance towards patient aggression.
Aggression and violence attitude | pre and post intervention
  Aggression and violence attitude was measured by the Management of Aggression and Violence Attitude Scale (MAVAS). The scale was consists of 7 items, rating from 1 (Strongly disagree) to 5 (Strongly agree). The sum of scores ranged from 7 to 35, with a higher score indicating a more positive attitude toward workplace violence.
Turnover Intentions | pre and post intervention
  Turnover Intentions was measured by the Turnover Intentions Scale (TIS). The scale was consists of 4 items, rating from 1 (Never) to 4 (Often). The sum of scores ranged from 4 to 16, with a higher score indicating a stronger turnover intention.

CONTACTS AND LOCATIONS:
Locations (1):
- TSGH, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma CY, Liao SJ, Chang YC, Chiang HH. Effectiveness of a theory-driven Brazilian jiu-jitsu-based medical self-defense training for nurses facing workplace violence: A multicenter quasi-experimental study. Int J Nurs Stud. 2026 Jan;173:105260. doi: 10.1016/j.ijnurstu.2025.105260. Epub 2025 Oct 22. PMID 41192105